CLINICAL TRIAL: NCT00051792
Title: Efficacy of Yoga for Self-Management of Dyspnea in COPD
Brief Title: Yoga for Treating Shortness of Breath in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT001168-01 (NIH)
Record Dates: First submitted 2003-01-16; First posted 2003-01-17 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Pulmonary Emphysema; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Pulmonary Emphysema; Bronchitis, Chronic | interventions — Yoga

INTERVENTIONS:
Behavioral: yoga

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of yoga in reducing shortness of breath in people with chronic obstructive pulmonary disease (COPD). Patients in this study must have moderate to severe COPD and be primarily limited by shortness of breath.

DETAILED DESCRIPTION:
Management of dyspnea (shortness of breath) is a major concern for patients with COPD. The efficacy of complementary exercises to manage dyspnea is unknown. Complementary exercises may be more congruent with patients' lifestyles and values than traditional exercise programs and can be adapted to changes in illness severity and disability. Yoga practice is a complementary therapy that people use to manage their dyspnea. The aims of this study are to: 1) develop a safe and feasible yoga program for patients with COPD; 2) test the efficacy of this program; and 3) determine whether physical performance, psychological well being, and health-related quality of life are positively affected by yoga practice.

Patients in this study will be randomized to receive yoga training or usual care for 12 weeks. Patients will be evaluated at study entry, after each session, and immediately after the training program.

ELIGIBILITY:
Inclusion criteria:

* Able to commit to a 12-week yoga class in San Francisco, California
* Moderate to severe COPD, clinically stable for at least 1 month prior to study entry
* Forced Expiratory Volume at one minute (FEV1) < 49% predicted after inhaled bronchodilator
* Activities of daily living limited by shortness of breath
* Ability to speak English and sign consent
* Patients receiving supplemental oxygen will be acceptable if their O2 saturation can be maintained at > 85% on < 6 L/min of nasal oxygen

Exclusion criteria:

* Symptomatic illness (e.g., cancer, left heart failure, ischemic heart disease, neuromuscular disease, psychiatric illness)
* Formal pulmonary rehabilitation training within 1 year prior to study entry

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-01; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Carrieri-Kohlman, RN, DNSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States